CLINICAL TRIAL: NCT03194802
Title: Efficacy of Sleeping Without Pills (SWOP), an Online Drug Tapering Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manitoba (Other)
Responsible Party: Principal Investigator, Dr. Nora Vincent, Clinical Psychologist, University of Manitoba
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H2017:066
Record Dates: First submitted 2017-06-19; First posted 2017-06-21 (Actual); Last update posted 2018-03-14 (Actual); Status verified 2018-03

CONDITIONS: Insomnia Chronic
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Sleep; Blood Glucose Self-Monitoring

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sleeping Without Pills Program (Experimental): Cognitive behavioral therapy; Motivational Interviewing; Scheduled and gradual drug tapering
  Interventions: Behavioral: Sleeping Without Pills Program
- Self-Monitoring (Active Comparator): Daily Self-monitoring of sleep and sleep medication using sleep diary
  Interventions: Behavioral: Self-monitoring

INTERVENTIONS:
Behavioral: Sleeping Without Pills Program — Participants receive this program online and are asked to log in daily for 6 weeks.
  Arms: Sleeping Without Pills Program
Behavioral: Self-monitoring — Participants enter sleep diary data online daily for 6 weeks
  Arms: Self-Monitoring

SUMMARY:
The aims of the study are to determine whether an online drug tapering program can lead to successful drug tapering in hypnotic dependent insomnia and whether such tapering is associated with improved daytime functioning and sleep.

DETAILED DESCRIPTION:
Insomnia is defined as difficulty with falling asleep, staying asleep, or early morning awakening. Chronic insomnia is estimated to affect 9-15% of the world's population. Lack of sleep increases a person's risk for many chronic diseases such as obesity, diabetes, cardiovascular disease, anxiety and depression. The two types of treatment available for chronic insomnia are cognitive behavioural therapy (CBT) and pharmacotherapy, the latter of which includes benzodiazepines and non-benzodiazepines.

The use of hypnotic medications is intended to be prescribed as a short-term treatment of one or two weeks, however this is not the case most of the time. Hypnotic abuse and dependency are prevalent issues that increase with advancing age. With the regular intake of these substances comes many adverse effects such as sedation, cognitive and psychomotor effects, falls and other accidents. Relative to non-drug users, cognitive events are 5.0 times more likely, psychomotor events are 3.0 times more likely, and daytime fatigue is 4.0 times more likely among drug users. Both non-benzodiazepines and benzodiazepines have the potential for dependency and withdrawal, although zolpidem and other non-benzodiazepine hypnotic agents have become the preferred drugs to manage insomnia due to the lower side effect profile. Withdrawal symptoms are associated with a rapid dose decrease or abrupt discontinuance of medication. These symptoms include rebound insomnia, anxiety, memory and concentration impairments and in severe states, psychotic symptoms, delirium and epileptic seizures.

A recent comparison of cost data associated with pharmacotherapy and cognitive behavioral therapy showed that CBT was significantly less costly than pharmacotherapy. Unfortunately, CBT is often not applied due to limited access to appropriately trained practitioners. The combination of equivalent efficacy, reduced costs, and favorable side-effect profile have made cognitive behavioural therapy (CBT) the preferred treatment for insomnia as evidenced by endorsements with the American Academy of Sleep Medicine. More recently, the delivery of CBT for insomnia has been enhanced to be provided through web-based portals. A number of web-based programs for insomnia have been developed with promising results. Some of these programs measured hypnotic use.

The effect size associated with online CBT (without drug tapering component) on reducing hypnotic drug use has been small, and these studies have employed a mix of participants, only some of whom are interested in tapering with variable levels of motivation. Studies comparing CBT plus drug tapering with drug tapering alone using booklets and in-person sessions have found that such interventions are moderately effective in reducing dosage and frequency of sleep medication usage.

The aims of the study are to determine whether an online drug tapering program (Sleeping without Pills; SWOP) can lead to successful drug tapering in hypnotic dependent insomnia (primary aim), and whether such tapering is associated with improved daytime functioning and sleep (secondary aims).

ELIGIBILITY:
Inclusion Criteria:

a) >= 18 years, b) access to high speed internet and computer, c) disturbance of sleep consisting of a delay in sleep onset, return to sleep or early morning awakening at least 3 nights/week for at least 3 months in duration, d) at least one symptom of daytime impairment, use of medication to promote sleep, e) use of medication to promote sleep (either <= 1mg lorazepam, <= .5mg clonazepam, <= 7.5mg zopiclone, <= 50 mg trazodone/amitriptyline, f) interested in medication tapering.

Exclusion Criteria:

a) shift work, b) head injury, c) acute crisis, d) seizure disorder, e) use of psychotropic drugs for problems other than sleep, f) use of medication interfering with sleep, g) recreational drug use, h) symptoms suggestive of alternative sleep disorder that is untreated, i) elevated use of alcohol (> 14 beverages/week for males, >12 beverages per week for females)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2017-06-05 (Actual); Primary Completion 2017-11-30 (Actual); Study Completion 2018-01-30 (Actual)

PRIMARY OUTCOMES:
Drug dose | 6 weeks
  Dose (mg) of sleep medication
Drug frequency | 6 weeks
  Frequency of use of sleep medication

SECONDARY OUTCOMES:
Dysfunctional Beliefs and Attitudes about Sleep Scale (DBAS) | 6 weeks
  maladaptive beliefs about sleep
Insomnia Severity Index | 6 weeks
  Concern about sleep and daytime impairment
Multi-Dimensional Fatigue Inventory | 6 weeks
  Daytime fatigue
Epworth Sleepiness Scale | 6 weeks
  Daytime sleepiness
Work and Social Adjustment Scale | 6 weeks
  Impact of sleep on work and living

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Health Psychology, Winnipeg, Manitoba, Canada